CLINICAL TRIAL: NCT06932692
Title: The BRAINMAP-DBS Study
Brief Title: The BRAINMAP-DBS Study: BRain Network AnalysIs usiNg 7-Tesla MRI and MAgnetoencephalograPhy for Deep Brain Stimulation
Acronym: BRAINMAP-DBS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Maarten Bot, MD, PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL86080.018.24; 10960102310022 (Other Grant/Funding Number: ZonMw Nationaal Plan Hoofdzaken); 09032232310059 (Other Grant/Funding Number: ZonMw Klinische Fellows)
Record Dates: First submitted 2025-04-10; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Deep Brain Stimulation; Parkinson Disease; Essential Tremor; Magnetoencephalography (MEG); MRI
Keywords: Deep Brain Stimulation; Parkinson's disease; Essential Tremor; 7 Tesla MRI; Magnetoencephalography; Brain networks
MeSH Terms: conditions — Parkinson Disease; Essential Tremor | interventions — Magnetoencephalography

STUDY DESIGN:
Intervention Model Description: Intervention: Patients with DBS for a minimum of six months will undergo an additional MEG scan. Application of 7T MRI for DBS is standard care and outcome scores used will be readily accessible from the already existing advanced electronic DBS database.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnetoencephalography (Other): Patients with DBS for a minimum of six months will undergo an additional MEG scan (intervention, for all participants). Application of 7T MRI for DBS is standard care and outcome scores used will be readily accessible from the already existing advanced electronic DBS database.
  Interventions: Other: magnetoencephalography

INTERVENTIONS:
Other: magnetoencephalography — 500 patients with Parkinson's disease and essential tremor will undergo magnetoencephalography

SUMMARY:
Rationale: Deep brain stimulation (DBS) is an effective treatment for essential tremor and Parkinson's disease. The effect of DBS relies on the modulation of dysfunctional motor brain networks and on average 50% motor improvement is achieved, using standardized motor evaluation scores. However, approximately 20% of treated patients show insufficient benefit, with less than 30% improvement. To improve outcomes through better electrode placement and selection of DBS electrical parameter programming, more advanced visualization of motor networks is needed; both anatomical (7-Tesla MRI) and functional (magnetoencephalography, MEG). Current DBS implantations are based on 1.5- or 3- Tesla MR scans. The resolution of these scans is not sufficient to visualize brain networks, preventing electrode placement directed at motor parts within the brain nucleus. In addition to the 7-Tesla MRI guided electrode placement, by applying MEG, programming will be directed at influencing the cortical motor areas, resulting in an overall decrease in dysfunctional network activity.

Objective: Primary objective of the study is to determine whether brain network visualization using 7T MRI and MEG improves motor symptoms as measured by the disease-specific Unified Parkinson's Disease Rating Scale (UPDRS-III) and Tremor Assessment Rating Scale (TETRAS); and quality of life as measured by the Parkinson's Disease Questionnaire 39 (PDQ-39). Secondary outcomes are: disease related daily functioning, adverse effects, operation time, quality of life (QUEST), patient satisfaction with treatment outcome and patient evaluation of treatment burden.

Study design: Single-center, prospective study with repeated measures; standardized assessments of motor skills and quality of life (UPDRS-III, TETRAS, PDQ-39) after DBS placement will be compared with scores after adjustments based on network analyses.

Study population: Enrollment will be ongoing from April 2024.

Intervention (if applicable): Patients with DBS for a minimum of six months will undergo an additional MEG scan. Application of 7T MRI for DBS is standard care and outcome scores used will be readily accessible from the already existing advanced electronic DBS database.

Main study parameters/endpoints: The co-primary outcome measures are the change in motor symptoms (measured by the UPDRS-III,TETRAS) and quality of life (measured by the PDQ-39). This is measured as part of standard care. The secondary outcome measures are the Amsterdam Linear Disability Score for functional health status, Starkstein apathy scale, Quality of Life Questionnaire in Essential Tremor (QUEST), patient satisfaction with the treatment, patient evaluation of treatment burden, operating time, hospitalization time, change of tremor medication, side effects and complications. The primary and secondary outcome scores are already stored in our advanced electronic DBS database.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The 7-Tesla MRI and MEG protocols (including stimulation parameters) already developed by our group and reported in (five) studies will be applied. After selecting the best DBS programming, the aim is to optimize DBS outcome by: a) increasing the mean improvement in motor function and quality of life by at least 10% and b) achieving a minimum of 30% improvement in motor function for each patient (measured by standardized assessment of motor function and quality of life). The proposed research project involves treatment options that are non-invasive and/or part of standard care in daily practice. The therapies will not be combined with other research products. Participation in this study constitutes negligible risk according to NFU criteria for human research.

DETAILED DESCRIPTION:
Deep brain stimulation for Parkinson's disease and essential tremor The effect of deep brain stimulation (DBS) relies on the modulation of dysfunctional motor brain networks.1,2 On average, 50% motor improvement is achieved, using standardized motor assessments. However, approximately 20% of patients shows insufficient benefit, with less than 30% improvement.3,4 To improve these outcomes, better electrode placement and selection of DBS electrical parameter programming is needed.5 This necessitates more advanced visualization of the intricate motor networks; both anatomical (7-Tesla MRI) and functional (MEG).11,12,13 Current DBS implantations are based on 1.5- or 3- Tesla MR scans. The resolution of these scans however, is not sufficient enough to visualize brain networks, preventing precise electrode placement directly at the motor parts within the small (size of a coffee bean) brain nucleus. In addition to the 7-Tesla MRI guided electrode placement, programming will be directed at influencing the cortical motor areas, by applying MEG, resulting in an overall decrease in dysfunctional network activity; instead of the "one-brain" model for everyone, DBS thereby becomes patient-specific, focused on one's own brain network.

Brain network analysis using 7-Tesla MRI and MEG The 7-Tesla MRI and MEG protocols already developed by our group and reported in (five) studies will be applied.6,7,8,9,10 In these studies we showed undistorted visualization of brain networks using 7-Tesla MRI and MEG in Parkinson disease patients that underwent DBS, and the potential to increase improvement in motor functioning by at least 10%. The 7-Tesla MRI network analysis, generated by combining T2 and diffusion weighted MRI, shows the (coloured) subdivisions of the brain nucleus and associated cortical projections. The MEG network analysis, generated from the MEG recordings, shows which cortical regions are affected (increase or decrease in activity, resulting in different colours) for each of the four individual electrode-contacts. Co-registration of the 7-Tesla MRI network, the MEG network and the CT scan will be performed for precise electrode localization. The result will show in which subdivision the DBS electrode-contact is located (placement), to which cortical area the subdivision projects and what activity patterns and changes therein are induced on the cortical areas (activation).16 Clinical test scores of the electrode-contact will then be correlated (regression analyses) with the network analysis. Since the entire network analysis will be visualized integrated on MRI, both individual analyses and group analyses (co-registration of networks of multiple patients) are possible, as well as application for the variable autoencoder. DBS location and programming based on 7-Tesla MRI and MEG network analysis will be used to optimize the outcome for beneficial clinical effects (suppression of tremor, bradykinesia, rigidity) with minimizing side effects (apathy, speech).15

For each patient, the total MEG recording will take 55 minutes. Nine short periods of unilateral stimulation will be performed with one of eight individual electrode-contacts, and one recording during DBS off in a randomized sequence. The effect of DBS on motor function (tremor, bradykinesia, rigidity, speech) is usually immediate and the assessment time is short (minutes). DBS settings can be temporarily adjusted during MEG recordings along with clinical assessment.

Upon completion of this process for all eight contacts of the electrode, the network analysis is performed and will show the DBS electrode-contact (left and right) which (solely) modulates the motor brain network. When the electrode-contact (DBS program) that the patient had before enrolment differs from the new 'brain network guided program' as determined by the network analysis, this new program is added to the DBS system. In the new program, margins for adjusting stimulation amplitude are set-up for later adjustments. The program that the patient had before enrolment in the study is kept as one of the programs on the device, which can be used as an 'escape option' by the patient if the newly programmed configurations have a worse clinical effect. After three months of network guided DBS standardized assessments of motor skills (UPDRS-III, TETRAS) will be performed as part of standard clinical care.

This project was set up in close collaboration with five DBS patients (patient-researchers). They identified regaining independence as the most important effect of DBS. They cited the possible adverse impact on cognition and mood (memory, speech, apathy) by DBS as their main concern. The discussed concerns were directly incorporated into the project.

Only few centers worldwide have a 7-Tesla MRI and MEG scan and therefore we will make this knowledge available through an open access database. We will apply the network analyses in the variable autoencoder (machine learning algorithm, a type of artificial intelligence) to generate prediction models with the help of the Department of Biomedical Engineering & Physics (Amsterdam UMC).14 The application of machine learning to large numbers of high-resolution scans allows for the generation of network models (connectomes) to indicate the most optimal location and programming for the DBS electrode; directly applicable for all DBS groups.

Feasibility Every patient undergoing DBS at the Amsterdam UMC undergoes a preoperative 7-Tesla MRI as part of standard care. In the 450 7-Tesla MR-scans we have performed to date, we rarely encountered non-compatible implants or severe claustrophobia. Every patient undergoes screening with a MRI safety questionnaire and MRI metal detector (preventing taking ferromagnetic materials into the MRI). 7-Tesla MRI is a non-invasive technique which causes no pain and, importantly, the electromagnetic fields produce no known tissue damage of any kind. The MR system may make loud tapping, knocking, or other noises at times during the procedure. Earplugs are provided to prevent problems that may be associated with noise generated by the scanner. At all times, the patient will be (visually) monitored and will be able to communicate with the 7-Tesla MRI technologist using an intercom system. The patient may (request to) stop the acquisition at any time by using the push button (hold by the patient continuously).

MEG recordings are non-invasive, pain free and have negligible risks. Based on literature and our own experience in 40 patients, MEG recordings during DBS are a safe procedure. Participants will make one extra trip to the MEG center located at location VUmc. Changing DBS settings within the limits stated in the individual DBS passport of the participants is a risk-free procedure. As participants are in supine position on a comfortable bed during MEG recordings, we do not expect them to experience unacceptable motor symptoms.

For the first time 7-Tesla MRI and MEG network analysis will be combined in in a large-scale prospective fashion; introducing patient specific network guided DBS electrode placement and programming.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, a subject must meet all of the following criteria:

* Age > 18 years;
* Idiopathic PD/ET with at least six months of DBS
* Underwent a preoperative 7-Tesla MRI scan

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Legally incompetent adults;
* No written informed consent.
* A spinal stimulation or deep brain stimulation system is not compatible with 7-Tesla MRI
* There a no implants inadmissible in the MEG, although patients will be questioned for possible (non-removable) implants such as pacemakerand/or dental as they may interfere with the magnetic signals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Essential Tremor Rating Assessment Scale (TETRAS) | assessment will be done before DBS and after 6 months of DBS
  The amount of decrease in motor symptoms indicated by change in the disease-specific Essential Tremor Rating Assessment Scale (TETRAS) after six months of deep brain stimulation. The TETRAS scores are between 0 and 64; higher scores indicating worse (more severe) tremor symptoms.
Unified Parkinson's Disease Rating Scale (UPDRS-III) | assessment will be done before DBS and after 6 months of DBS
  The amount of decrease in motor symptoms indicated by change in the disease-specific Unified Parkinson's Disease Rating Scale (UPDRS-III) after six months of deep brain stimulation. The UPDRS-III scores are between 7 and 86; higher scores indicating worse (more severe) motor symptoms.
Parkinson's disease questionnaire-39 | assessment will be done before DBS and after 6 months of DBS
  The Parkinson's Disease Questionnaire (PDQ-39) assesses how often people with Parkinson's experience difficulties across 8 dimensions of daily living including relationships, social situations and communication. It also assesses the impact of Parkinson's on specific dimensions of functioning and wellbeing. The scores are between 0 and 100 (the sum of all 39 items), higher score indicating more health problems.

SECONDARY OUTCOMES:
The Amsterdam Linear Disability Score for functional health status | assessment will be done before DBS and after 6 months of DBS
  The Amsterdam Linear Disability Score (ALDS) is a generic itembank which measures disability, as expressed by the ability to perform activities of daily living. These scores are linearly transformed into values between 0 and 100. Lower scores indicate more disability.
Starkstein apathy scale | assessment will be done before DBS and after 6 months of DBS
  The 14-item Starkstein Apathy Scale (SAS) is used to measure the severity of apathetic symptoms in Parkinson disease. The scores are between 0 and 42. Higher scores indicating worse apathy.
Quality of Life in Essential Tremor Questionnaire | assessment will be done before DBS and after 6 months of DBS
  The Quality of Life in Essential Tremor Questionnaire (QUEST) is a 30-item scale developed specifically for patients with essential tremor to measure items impacting perceived quality of life (QOL) that generic QOL measures do not effectively capture, including activities of daily living that are affected by essential tremor. The QUEST was made to be relatively brief and easy for patients to use.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
We will develop a prediction model based on the generated networks (connectomes) using the variable autoencoder (machine learning algorithm). Create a (7-Tesla MRI and MEG) open access database including the connectomes; applicable in any center for both clinical and fundamental studies.
  This database will not show traceable individual participant data

REFERENCES:
- [Background] Boon LI, Hillebrand A, Potters WV, de Bie RMA, Prent N, Bot M, Schuurman PR, Stam CJ, van Rootselaar AF, Berendse HW. Motor effects of deep brain stimulation correlate with increased functional connectivity in Parkinson's disease: An MEG study. Neuroimage Clin. 2020;26:102225. doi: 10.1016/j.nicl.2020.102225. Epub 2020 Feb 21. PMID 32120294
- [Background] Boon LI, Potters WV, Hillebrand A, de Bie RMA, Bot M, Richard Schuurman P, van den Munckhof P, Twisk JW, Stam CJ, Berendse HW, van Rootselaar AF. Magnetoencephalography to measure the effect of contact point-specific deep brain stimulation in Parkinson's disease: A proof of concept study. Neuroimage Clin. 2023;38:103431. doi: 10.1016/j.nicl.2023.103431. Epub 2023 May 10. PMID 37187041
- [Background] Zoon TJC, Mathiopoulou V, van Rooijen G, van den Munckhof P, Denys DAJP, Schuurman PR, de Bie RMA, Bot M. Apathy following deep brain stimulation in Parkinson's disease visualized by 7-Tesla MRI subthalamic network analysis. Brain Stimul. 2023 Sep-Oct;16(5):1289-1291. doi: 10.1016/j.brs.2023.08.013. Epub 2023 Aug 22. PMID 37619890
- [Background] Mathiopoulou V, Rijks N, Caan MWA, Liebrand LC, Ferreira F, de Bie RMA, van den Munckhof P, Schuurman PR, Bot M. Utilizing 7-Tesla Subthalamic Nucleus Connectivity in Deep Brain Stimulation for Parkinson Disease. Neuromodulation. 2023 Feb;26(2):333-339. doi: 10.1016/j.neurom.2022.01.003. Epub 2022 Feb 23. PMID 35216874
- [Background] Verlaat L, Rijks N, Dilai J, Admiraal M, Beudel M, de Bie RMA, van der Zwaag W, Schuurman R, van den Munckhof P, Bot M. 7-Tesla Magnetic Resonance Imaging Scanning in Deep Brain Stimulation for Parkinson's Disease: Improving Visualization of the Dorsolateral Subthalamic Nucleus. Mov Disord Clin Pract. 2024 Apr;11(4):373-380. doi: 10.1002/mdc3.13982. Epub 2024 Feb 22. PMID 38385792